CLINICAL TRIAL: NCT03976752
Title: Body Compartment Pharmacokinetics of Anti-retroviral Agents That May be Considered for Future On-demand Peri-exposure HIV Prophylaxis Regimens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen Kelley, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB00108386
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: HIV/AIDS
Keywords: HIV; MSM; Anti-retrovirals; Pharmacokinetics; Peri-exposure HIV prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pre-drug (No Intervention): Participants enrolled in the pre-drug arm will not receive any drug. At visit 2, they will undergo blood, urine, penile swab, cheek swab, rectal swab and rectal biopsy collection.
- Genvoya - 2 and 48 hours specimen collection (Experimental): Specimen collection 2 hours after taking the medication in the clinic (visit 4), and 48 hours after taking the medication in the clinic (visit 5).
  Interventions: Drug: Genvoya
- Genvoya - 4 and 72 hours specimen collection (Experimental): Specimen collection 4 hours after taking the medication in the clinic (visit 4), and 72 hours after taking the medication in the clinic (visit 5).
  Interventions: Drug: Genvoya
- Genvoya - 24 and 96 hours specimen collection (Experimental): Specimen collection 24 hours after taking the medication in the clinic (visit 4), and 96 hours after taking the medication in the clinic (visit 5).
  Interventions: Drug: Genvoya
- Genvoya - Single time point specimen collection (Experimental): Specimen collection 8 hours after taking the medication in the clinic (visit 4).
  Interventions: Drug: Genvoya

INTERVENTIONS:
Drug: Genvoya — Genvoya is a fixed-dose combination anti-retroviral drug containing tenofovir alafenamide (TAF), emtricitabine (FTC), elvitegravir (EVG), and cobicistat.
  At the second study visit, participants will be provided with a single dose of Genvoya, and instructed to take the dose at home with documentation by digital, time-stamped photo or video. At the third study visit, which will occur 24 hours after home dosing, participants will be given another single dose of Genvoya at the clinic.
  Other Names: Cobicistat/Elvitegravir/Emtricitabine/Tenofovir alafenamide
  Arms: Genvoya - 2 and 48 hours specimen collection; Genvoya - 24 and 96 hours specimen collection; Genvoya - 4 and 72 hours specimen collection; Genvoya - Single time point specimen collection

SUMMARY:
This study is being conducted to determine if the uptake of anti-HIV medication, called Genvoya®, at different time-frames, is different at several body sites, including mucosal tissues. This medication might be considered for on-demand PEP regimens in the future.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) continue to be disproportionately affected by HIV. The majority of MSM acquire HIV after exposure to the rectal mucosa through unprotected receptive anal intercourse. Post-exposure-prophylaxis (PEP) is an intervention that is used to prevent HIV infection soon (72 hours) after a potential exposure. HIV-negative people with a possible exposure to HIV are instructed to take 28 days of a combination anti-HIV medication regimen, Truvada® + Raltegravir.

This study is being conducted to determine if the uptake of another anti-HIV medication, called Genvoya®, at different time-frames, is different at several body sites, including mucosal tissues. This medication might be considered for on-demand PEP regimens in the future.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-negative man who reports receptive anal sex with another man in the last 6 months
2. Aged 18-49 years
3. Not currently taking PrEP and no plans to initiate during study
4. Not currently taking PEP
5. Able to provide informed consent in English
6. No plans for relocation in the next 3 months
7. Willing to undergo peripheral blood, penile swabs, urine, and rectal biopsy sampling
8. Willing to use study products as directed
9. Willing to abstain from receptive anal intercourse 3 days prior to starting study product and for the duration of the study and for 7 days after any rectal biopsy procedure.
10. Hepatitis B surface antigen (HBsAg) must be negative (screening lab test)
11. Creatine clearance >60 ml/min

Exclusion Criteria:

1. History of inflammatory bowel disease or other inflammatory, infiltrative, infectious or vascular condition involving the lower gastrointestinal tract that, in the judgment of the investigators, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel
2. Currently infected with hepatitis virus and/ or have liver disease
3. Current or chronic history of kidney disease
4. Significant laboratory abnormalities at baseline visit, including but not limited to:

   1. Hgb ≤ 10 g/dL
   2. Partial thromboplastin time (PTT) > 1.5x upper limit of normal (ULN) or international normalized ratio (INR) > 1.5x ULN
   3. Platelet count <100,000
   4. Creatinine clearance <60
   5. HBsAg reactive
5. Any known medical condition that, in the judgment of the investigators, increases the risk of local or systemic complications of endoscopic procedures or pelvic examination, including but not limited to:

   1. Uncontrolled or severe cardiac arrhythmia
   2. Recent major abdominal, cardiothoracic, or neurological surgery
   3. History of uncontrolled bleeding diathesis
   4. History of colonic, rectal, or vaginal perforation, fistula, or malignancy
   5. History or evidence on clinical examination of ulcerative, suppurative, or proliferative lesions of the anorectal mucosa, or untreated sexually transmitted disease with mucosal involvement
6. Continued need for, or use during the 14 days prior to enrollment, of the following medications:

   1. Aspirin or more than 4 doses of NSAIDs
   2. Warfarin, heparin (low-molecular weight or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
   3. Any form of rectally administered agent besides lubricants or douching used for sexual intercourse
7. Continued need for, or use during the 90 days prior to enrollment, of the following medications:

   1. Systemic immunomodulatory agents
   2. Supraphysiologic doses of steroids (short course steroids less than 7 days duration, allowable at the discretion of the investigators)
   3. Experimental medications, vaccines, or biologicals
8. Intent to use HIV antiretroviral pre/post-exposure prophylaxis (PrEP or PEP) during the study, outside of the study procedures
9. Symptoms of an untreated rectal sexually transmitted infection (e.g. rectal pain, discharge, bleeding, etc.)
10. Current use of hormonal therapy
11. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
12. Participants taking potent inhibitors (e.g. itraconazole, diltiazem) or inducers (e.g. rifampin, phenytoin) of the CYP3A4 enzyme that also metabolizes Genvoya will be excluded from the study

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 41 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (e.g., text, tables, figures, and appendices), will be available. The study protocol will be available. Data will become available Beginning 9 months and ending at 36 months following publication to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Data will become available beginning 9 months and ending at 36 months following article publication.
Access Criteria: Proposals should be directed to colleen.kelley@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Hope Clinic in Atlanta, Georgia, USA. Participant enrollment began on March 13, 2019 and all follow up was completed September 20, 2019.
Pre-assignment Details: After the completion of enrollment in the Pre-drug arm, enrollment began sequentially in Arm A, followed by Arm B and Arm C. Arms A, B, and C were further broken down into two different sub-groups, determining the timing of the rectal swab and biopsy procedure. Arm D was enrolled last and included a single time point specimen collection. Participants were able to take part in more than one study arm, with at least a 6 week period after completion of one study arm before beginning another one.
Groups:
- Genvoya: Genvoya is a fixed-dose combination anti-retroviral drug containing tenofovir alafenamide (TAF), emtricitabine (FTC), elvitegravir (EVG), and cobicistat. At the second study visit, participants will be provided with a single dose of Genvoya, and instructed to take the dose at home with documentation by digital, time-stamped photo or video. At the third study visit, which will occur 24 hours after home dosing, participants will be given another single dose of Genvoya at the clinic.
  Participants took Genvoya and had specimens collected at different time points.
  * Arm A: specimen collection occurred 2 hours and after taking the medication in the clinic (visit 4), and 48 hours after taking the medication in the clinic (visit 5)
  * Arm B: specimen collection occurred 4 hours and after taking the medication in the clinic (visit 4), and 72 hours after taking the medication in the clinic (visit 5)
  * Arm C: specimen collection occurred 24 hours and after taking the medication in the clinic (visit 4), and 96 hours after taking the medication in the clinic (visit 5)
  * Arm D: specimen collection occurred 8 hours after taking the medication in the clinic (visit 4), for a single time point of specimen collection
Period: Overall Study
Arm/Group | Pre-drug | Genvoya
Started | 4 | 37
Started Study Arm A | 0 | 14
Completed Study Arm A | 0 | 8
Started Study Arm B | 0 | 8
Completed Study Arm B | 0 | 8
Started Study Arm C | 0 | 11
Completed Study Arm C | 0 | 8
Started Study Arm D | 0 | 6
Completed Study Arm D | 0 | 4
Completed | 3 | 28
Not Completed | 1 | 9

BASELINE CHARACTERISTICS:
Groups:
- Pre-drug: Participants enrolled in the pre-drug arm did not receive any drug. At visit 2, they underwent blood, urine, penile swab, cheek swab, rectal swab and rectal biopsy collection.
- Genvoya: Genvoya is a fixed-dose combination anti-retroviral drug containing tenofovir alafenamide (TAF), emtricitabine (FTC), elvitegravir (EVG), and cobicistat. At the second study visit, participants will be provided with a single dose of Genvoya, and instructed to take the dose at home with documentation by digital, time-stamped photo or video. At the third study visit, which will occur 24 hours after home dosing, participants will be given another single dose of Genvoya at the clinic.
  Participants took Genvoya and had specimens collected at different time points. Arm A: specimen collection occurred 2 hours and after taking the medication in the clinic (visit 4), and 48 hours after taking the medication in the clinic (visit 5) Arm B: specimen collection occurred 4 hours and after taking the medication in the clinic (visit 4), and 72 hours after taking the medication in the clinic (visit 5) Arm C: specimen collection occurred 24 hours and after taking the medication in the clinic (visit 4), and 96 hours after taking the medication in the clinic (visit 5) Arm D: specimen collection occurred 8 hours after taking the medication in the clinic (visit 4), for a single time point of specimen collection
- Total: Total of all reporting groups
Arm/Group | Pre-drug | Genvoya | Total
Number analyzed (Participants) | 4 | 37 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 4 | 36 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 37 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 26 | 30
  White | 0 | 7 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 37 | 41

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Tenofovir (TFV)
Description: Median drug concentrations of the TFV component of Genvoya were determined at baseline and at each of the protocol specified follow-up time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: Data are reported per intervention, based on the time points of sample collection for each study arm (two participants were in multiple study arms). Analysis of drug concentrations in participants in the Pre-drug arm was not performed as no drugs were administered to this study arm.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng/mL
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 0 [0 to 0] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 0 [0 to 0] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 0 [0 to 0]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 0 [0 to 13] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 0 [0 to 0] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 0 [0 to 0] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 0 [0 to 60] |

2. Primary Outcome: Plasma Concentration of Emtricitabine (FTC)
Description: Median drug concentrations of the FTC component of Genvoya were determined at baseline and at each of the protocol specified follow-up time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng/mL
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 2710 [1765 to 3345] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 1725 [747 to 2565] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 300 [225 to 351]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 113 [37 to 258] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 0 [0 to 768] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 0 [0 to 0] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 0 [0 to 107] |

3. Primary Outcome: Plasma Concentration of Elvitegravir (EVG)
Description: Median drug concentrations of the EVG component of Genvoya were determined at baseline and at each of the protocol specified follow-up time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng/mL
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 2243 [916 to 3455] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 1818 [1230 to 4095] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 283 [105 to 421]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 232 [22 to 527] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 0 [0 to 69] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 0 [0 to 0] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 0 [0 to 18] |

4. Secondary Outcome: Peripheral Blood Mononuclear Cell (PBMC) Concentration of Tenofovir-diphosphate (TFV-DP)
Description: A peripheral blood mononuclear cell (PBMC) is any peripheral blood cell having a round nucleus: lymphocytes (T cells, B cells, natural killer (NK) cells) and monocytes. Median drug concentrations were determined at baseline and at each of the protocol specified follow-up time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: fmol/10^6 cells
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
fmol/10^6 cells
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 569 [262 to 1287] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 621 [156 to 1375] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 375 [270 to 1294]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 429 [276 to 659] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 291 [202 to 421] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 158 [81 to 436] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 117 [92 to 227] |

5. Secondary Outcome: Peripheral Blood Mononuclear Cell (PBMC) Concentration of Emtricitabine-triphosphate (FTC-TP)
Description: A peripheral blood mononuclear cell (PBMC) is any peripheral blood cell having a round nucleus: lymphocytes (T cells, B cells, NK cells) and monocytes. Median drug levels were determined at baseline and at each of the protocol specified follow-up time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: fmol/10^6 cells
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
fmol/10^6 cells
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 7705 [5230 to 8750] |  |  |
  4 hour: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hour |  | 7800 [3200 to 11650] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 6855 [5380 to 7710]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 5140 [3110 to 7740] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 2120 [1517 to 3390] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 955 [648 to 2210] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 714 [333 to 6000] |

6. Other Pre Specified Outcome: Rectal Tissue Concentration of Tenofovir (TFN)
Description: Median drug concentrations in rectal tissue of the TFN component of Genvoya were determined at baseline and at each of the protocol specified time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mg
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng/mg
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 0 [0 to 0.48] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 0.30 [0 to 1.23] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 0.01 [0 to 0.01]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 0.03 [0 to 1.20] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 0 [0 to 0] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 0 [0 to 0] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 0 [0 to 0] |

7. Other Pre Specified Outcome: Rectal Tissue Concentration of Emtricitabine (FTC)
Description: Median drug concentrations in rectal tissue of the FTC component of Genvoya were determined at baseline and at each of the protocol specified time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mg
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng/mg
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 9.54 [6.23 to 10.43] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 9.25 [0 to 12.11] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 0.17 [0.11 to 0.19]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 1.23 [0.29 to 12.86] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 0.02 [0 to 4.93] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 0 [0 to 0] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 0.02 [0.02 to 0.03] |

8. Other Pre Specified Outcome: Rectal Tissue Concentration of Elvitegravir (EVG)
Description: Median drug concentrations in rectal tissue of the EVG component of Genvoya were determined at baseline and at each of the protocol specified time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mg
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng/mg
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 51.23 [28.19 to 69.04] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 41.47 [8.95 to 66.17] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 0.31 [0.05 to 0.51]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 0.60 [0.29 to 40.02] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 1.03 [0 to 2.46] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 0 [0 to 0] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 0.02 [0.02 to 0.03] |

9. Other Pre Specified Outcome: Rectal Tissue Concentration of Tenofovir-diphosphate (TFV-DP)
Description: Median drug concentrations of TFV-DP in rectal tissue were determined at baseline and at each of the protocol specified follow-up time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: fmol/mg
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
fmol/mg
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 39.1 [34.2 to 74.6] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 45.9 [15.7 to 135.4] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 23.7 [14.7 to 27.4]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 20.2 [5.0 to 35.7] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 18.2 [15.9 to 22.1] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 11.9 [6.7 to 22.2] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 14.7 [4.6 to 1926.0] |

10. Other Pre Specified Outcome: Rectal Tissue Concentration of Emtricitabine-triphosphate (FTC-TP)
Description: Median drug concentrations of FTC-TP in rectal tissue were determined at baseline and at each of the protocol specified follow-up time points. Concentrations below the limit of quantification (LOQ) are assigned a value of zero.
Time Frame: Baseline, and 2, 4, 8, 24, 48, 72, 96 hours after taking the second dose of medication
Population: as for outcome 1
Measure: Median (Full Range); unit: fmol/mg
Arm/Group | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
Number analyzed (Participants) | 8 | 8 | 8 | 4
fmol/mg
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  2 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  2 hours | 187.5 [146.6 to 255.9] |  |  |
  4 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  4 hours |  | 198.2 [68.9 to 365.8] |  |
  8 hours: number analyzed (Participants) | 0 | 0 | 0 | 4
  8 hours |  |  |  | 116.5 [62.3 to 176.6]
  24 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  24 hours |  |  | 104.3 [19.5 to 184.5] |
  48 hours: number analyzed (Participants) | 8 | 0 | 0 | 0
  48 hours | 56.3 [18.1 to 91.7] |  |  |
  72 hours: number analyzed (Participants) | 0 | 8 | 0 | 0
  72 hours |  | 15.1 [7.3 to 52.3] |  |
  96 hours: number analyzed (Participants) | 0 | 0 | 8 | 0
  96 hours |  |  | 12.5 [6.3 to 141.3] |

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected from the time of study enrollment, at the screening visit, through two days after the biopsy (up to seven weeks total).
Description: Adverse events are reported per intervention (two participants were in multiple study arms).
Groups:
- Genvoya - 2 and 48 Hours Specimen Collection: Specimen collection 2 hours after taking the medication in the clinic (visit 4), and 48 hours after taking the medication in the clinic (visit 5).
  Genvoya: Genvoya is a fixed-dose combination anti-retroviral drug containing tenofovir alafenamide (TAF), emtricitabine (FTC), elvitegravir (EVG), and cobicistat.
  At the second study visit, participants will be provided with a single dose of Genvoya, and instructed to take the dose at home with documentation by digital, time-stamped photo or video. At the third study visit, which will occur 24 hours after home dosing, participants will be given another single dose of Genvoya at the clinic.
- Genvoya - 4 and 72 Hours Specimen Collection: Specimen collection 4 hours after taking the medication in the clinic (visit 4), and 72 hours after taking the medication in the clinic (visit 5).
  Genvoya: Genvoya is a fixed-dose combination anti-retroviral drug containing tenofovir alafenamide (TAF), emtricitabine (FTC), elvitegravir (EVG), and cobicistat.
  At the second study visit, participants will be provided with a single dose of Genvoya, and instructed to take the dose at home with documentation by digital, time-stamped photo or video. At the third study visit, which will occur 24 hours after home dosing, participants will be given another single dose of Genvoya at the clinic.
- Genvoya - 24 and 96 Hours Specimen Collection: Specimen collection 24 hours after taking the medication in the clinic (visit 4), and 96 hours after taking the medication in the clinic (visit 5).
  Genvoya: Genvoya is a fixed-dose combination anti-retroviral drug containing tenofovir alafenamide (TAF), emtricitabine (FTC), elvitegravir (EVG), and cobicistat.
  At the second study visit, participants will be provided with a single dose of Genvoya, and instructed to take the dose at home with documentation by digital, time-stamped photo or video. At the third study visit, which will occur 24 hours after home dosing, participants will be given another single dose of Genvoya at the clinic.
- Genvoya - Single Time Point Specimen Collection: Specimen collection 8 hours after taking the medication in the clinic (visit 4).
  Genvoya: Genvoya is a fixed-dose combination anti-retroviral drug containing tenofovir alafenamide (TAF), emtricitabine (FTC), elvitegravir (EVG), and cobicistat.
  At the second study visit, participants will be provided with a single dose of Genvoya, and instructed to take the dose at home with documentation by digital, time-stamped photo or video. At the third study visit, which will occur 24 hours after home dosing, participants will be given another single dose of Genvoya at the clinic.
Arm/Group | Pre-drug | Genvoya - 2 and 48 Hours Specimen Collection | Genvoya - 4 and 72 Hours Specimen Collection | Genvoya - 24 and 96 Hours Specimen Collection | Genvoya - Single Time Point Specimen Collection
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/14 | 0/8 | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/14 | 0/8 | 0/11 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/14 | 0/8 | 0/11 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03976752/Prot_SAP_000.pdf